CLINICAL TRIAL: NCT01145469
Title: Genome Wide Association Study Evaluating Genetic Factors Related to the Efficacy and Tolerability of Fludarabine Treatment in Patients With CLL
Brief Title: Biomarkers in DNA Samples From Patients With Chronic Lymphocytic Leukemia Previously Treated With Fludarabine-Based Therapy
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000674957; ECOG-E2997T2
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of DNA in the laboratory from patients who received fludarabine-based treatment may help doctors learn more about the effects of fludarabine on cells. It may also help doctors understand how well patients respond to treatment.

PURPOSE: This research study is studying DNA samples from patients with chronic lymphocytic leukemia previously treated with fludarabine-based therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify genetic characteristics associated with the efficacy and toxicity of fludarabine-based treatment in patients with chronic lymphocytic leukemia who participated on E2997.
* To validate these genetic characteristics with a cancer cell model system to confirm association and dissect the mechanism of effect.

OUTLINE: Archived DNA samples are analyzed for genetic characteristics associated with the efficacy and toxicity to fludarabine-based treatment using Affymetrix 6.0 single nucleotide polymorphism arrays. The results are then compared with data of genes identified in a cancer cell model system, and with clinical data (response, toxicity, overall survival, and progression-free survival) associated with each patient sample.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia
* Archived DNA samples
* Received fludarabine with versus without cyclophosphamide on clinical trial E2997

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E4402 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-01 (Actual)

PRIMARY OUTCOMES:
Association of single SNP genotype with overall and progression-free survival | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Tait D. Shanafelt, MD, Principal Investigator — Mayo Clinic